CLINICAL TRIAL: NCT03618576
Title: Effectiveness of the Computerized Balance Rehabilitation After Hip Fracture Surgery
Brief Title: Balance Rehabilitation After Hip Fracture Surgery
Acronym: BRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Yoon Lee, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-2018-46
Record Dates: First submitted 2018-07-19; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance exercise group (Experimental): During the 2-week postoperative intervention period, patients will participate in the hospital's exercise program beginning 5-7 days after HFS. All participants will follow the computer-based balance specific exercise (BSE) program.
  Interventions: Procedure: Balance specific exercise

INTERVENTIONS:
Procedure: Balance specific exercise — Balance specific exercise consists of total 10 days' physical therapy (PT) sessions (twice per day for 60 min) after surgery. It will be conducted with a computed posturographic system for diagnostics of balance and movement skills (Balance Master® System NeuroCom®) designed to objectively quantify balance and postural function of different origin. PT (weight-bearing, strengthening, gait training, aerobic, and functional exercises) was gradually increased based on the patient's functional level. Intensive patient education by multidisciplinary rehabilitation members was also provided.

SUMMARY:
The overall functional gain by balance rehabilitation after hip fracture surgery has not yet been fully investigated. Therefore, clinical studies should be conducted to evaluate the effectiveness of systematic and safe balance rehabilitation in patients after hip fracture. Investigators aim to evaluate the effect of computer-based balance specific exercise on the performance and balance ability of the elderly women who underwent hip fracture surgery. Investigators also investigate the intervention can reduce their fear of falling and coping ability. This study was designed as a prospective, open-label, single-center trial at a tertiary hospital setting. During the 2-week postoperative intervention period, patients will participate in the hospital's exercise program beginning 5-7 days after hip fracture surgery. All participants will follow the computer-based balance specific exercise program. Functional outcomes will be measure periodically for 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elderly female patients (≥ 65 years old) who have undergone surgery for femoral neck, intertrochanteric, or subtrochanteric fracture, regardless of surgery type (internal fixation, bipolar hemiarthroplasty, or total hip arthroplasty)

Exclusion Criteria:

* 1) hip surgery for infection, arthritis, implant loosening, or avascular necrosis;
* 2) femoral shaft fracture, acetabular fracture, isolated fracture of the greater or lesser tuberosity, or periprosthetic fracture;
* 3) pathologic fracture;
* 4) combined multiple fracture;
* 5) revision surgery;
* 6) severe cognitive dysfunction (obey command ≤ 1 step);
* 7) cannot stand by supporting a fixed walker at 5 days after operation;
* 8) patients who refuse to participate in a clinical trial

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change of Berg balance scale | Change from Baseline Berg balance scale at 6 months
  Berg balance scale (total score; 0 to 56)

SECONDARY OUTCOMES:
Functional Ambulatory Category | Before intervention, After 2 weeks' intervention, 3 and 6 months after surgery
  Functional Ambulatory Category (categorical score; 0 to 5)
Functional Independence Measure: locomotion | Before intervention, After 2 weeks' intervention, 3 and 6 months after surgery
  Functional Independence Measure (subscale of locomotion: 1 to 7)
Modified falls efficacy scale | Before intervention, After 2 weeks' intervention, 3 and 6 months after surgery
  Modified falls efficacy scale (total score: 0 to 140)
Presence of Fear of falling | Before intervention, After 2 weeks' intervention, 3 and 6 months after surgery
  Fear of falling (yes or no; by simple question "Are you afraid of falling?")
Modified Barthel index | Before intervention, After 2 weeks' intervention, 3 and 6 months after surgery
  Modified Barthel index (tota; score: 0 to 100)
Short physical performance scale | Before intervention, After 2 weeks' intervention, 3 and 6 months after surgery
  Short physical performance scale (total score: 0 to 12)

IPD SHARING:
Plan to Share IPD: No